CLINICAL TRIAL: NCT03401632
Title: Enteral Nutrition in Critically Ill Patients Undergoing Vasoactive Drugs Therapy. The NUTRIVAD Study.
Brief Title: Enteral Nutrition and Vasoactive Drugs
Acronym: NUTRIVAD
Status: Completed | Type: Observational
Sponsor: Hospital Severo Ochoa (Other)
Collaborators: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Principal Investigator, Jose Luis Flordelis Lasierra, MD, PhD, Principal Investigator, Hospital Severo Ochoa
Other Study IDs: HSeveroOchoa
Record Dates: First submitted 2018-01-03; First posted 2018-01-17 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Enteral Nutrition; Vasopressor Agents; Hemodynamics Instability; Critical Care
Keywords: Enteral nutrition; Vasoactive Drugs; Critical Care
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Enteral nutrition — Enteral nutrition support

SUMMARY:
Enteral nutrition in critically ill patients undergoing vasoactive support due to hemodynamic instability is controversial. Hypothesis: enteral nutrition delivered in such patients can be feasible and safe.

DETAILED DESCRIPTION:
Nutrition support in critically ill patients undergoing vasoactive support due to hemodynamic instability is controversial and challenging. However, if it is delivered according to an enteral nutrition protocol and under proper medical supervision, it can be feasible and safe. The present multicenter prospective study was designed to examine the feasibility and safety of enteral nutrition support in such patients.

ELIGIBILITY:
Inclusion Criteria:

* Authorization to participate in the study by informed consent.
* Dependence of vasoactive drugs and/or mechanical circulatory support to at least 48 hours from Intensive Care Unit admission.
* Invasive mechanical ventilation time of at least 48 hours.
* Expected survival greater than 72 hours.
* ICU Stay greater than or equal to 72 hours.

Exclusion Criteria:

* Refusal to participate in the study.
* Refractory shock, defined as the progressive elevation of the dose of vasoactive drugs and / or markers of tissue hypoperfusion, or mean arterial pressure ≤ 60 mm Hg despite the therapeutic maneuvers.
* History of significant abdominal vascular disease (ischemic colitis, chronic mesenteric ischemia, aortic aneurysm abdominal, aortic dissection with involvement of mesenteric vessels, etc).
* Absolute contraindication for the onset of enteral nutrition (active gastrointestinal hemorrhage, intestinal obstruction, etc.) or patients with a non-functional gastrointestinal tract.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adults.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-01-15 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Dose of vasoactive drugs. | Daily to a maximum of 14 days after Intensive Care Unit Admission.
  Dose of vasoactive drugs (highest daily), in μg/kg/min.
Kilocalories delivered by enteral route and Energy balance (Kilocalories delivered by enteral nutrition - (minus) enteral nutrition target in Kilocalories). | Daily to a maximum of 14 days after Intensive Care Unit Admission.
  Main Enteral nutrition efficacy-related variables. Enteral nutrition target was 25 Kilocalories/Kg, if body mass index (BMI) was between 20 and 30. Corrections were made if BMI was under 20/ or over 30.
Enteral nutrition-related mesenteric ischemia. | Daily to a maximum of 14 days after Intensive Care Unit Admission.
  Main enteral nutrition- safety related variable, suspected by the presence of warning signs (clinical, analytical, radiological), confirmed by laparotomy/laparoscopy, arteriography or angio-CT.

SECONDARY OUTCOMES:
Blood lactate. | Daily to a maximum of 14 days after Intensive Care Unit Admission.
  Daily peak blood lactate, in mmol/l.
Cardiac index. | Daily to a maximum of 14 days after Intensive Care Unit Admission.
  Daily lowest cardiac index, in L/min/m^2
Mechanical circulatory support. | Daily to a maximum of 14 days after Intensive Care Unit Admission.
  Dependence on Mechanical circulatory support (intra-aortic balloon pump, mechanical circulatory assistance, or extracorporeal membrane oxygenation).
Time from Intensive Care Unit admission to the start of enteral nutrition. | Up to 120 hours after Intensive Care Unit Admission.
  Time frame in hours from Intensive Care Unit admission to the start of enteral nutrition.
Nutrition Tolerance. | Daily to a maximum of 14 days after Intensive Care Unit Admission.
  Kilocalories delivered by enteral nutrition, divided by nutrition target in Kilocalories, expressed as percentage.
High gastric residual volume. | Daily to a maximum of 14 days after Intensive Care Unit Admission
  Gastric residual volume was described as high when >500 mL was obtained in each assessment.
Abdominal distention. | Daily to a maximum of 14 days after Intensive Care Unit Admission.
  A change in the abdomen detected in a physical examination, with an increase in abdominal cavity size relative to that recorded in the pre-enteral nutrition examination
Regurgitation. | Daily to a maximum of 14 days after Intensive Care Unit Admission.
  Presence of Enteral nutrition feed in the oral cavity or oropharynx, as well as its spontaneous drainage by the oral and/or nasal route
Enteral nutrition-related diarrhea. | Daily to a maximum of 14 days after Intensive Care Unit Admission.
  5 or more liquid stools in 24 hours or more than two 1000-mL stool volumes, each deposited over a 24-hour period.
Constipation. | Daily to a maximum of 14 days after Intensive Care Unit Admission.
  Lack of bowel movements in 7 days from the onset of enteral nutrition or for 3 days in the first week of admission.
Bronchoaspiration. | Daily to a maximum of 14 days after Intensive Care Unit Admission.
  The presence of respiratory secretions of similar characteristics to the prescribed enteral nutrition feed, confirmed by the glucose-oxidase technique in tracheal secretion.
Nasogastric tube complications. | Daily to a maximum of 14 days after Intensive Care Unit Admission.
  Obstruction or misplacement/accidental extubation.
Enteral nutrition interruptions. | Daily to a maximum of 14 days after Intensive Care Unit Admission.
  Need to interrupt or discontinue enteral nutrition (and reasons)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luis Flordelís Lasierra, MD, PhD, Study Director — Hospital Universitario Severo Ochoa. Leganés. Madrid. Spain.; Juan Carlos Montejo González, MD, PhD, Study Chair — Hospital Universitario 12 de Octubre. Madrid. Spain; Luis Juan Terceros Almanza, MD, Principal Investigator — Hospital Universitario 12 de Octubre. Madrid. Spain; Antonio Luis Blesa Malpica, MD, PhD, Principal Investigator — Hospital Universitario Clínico San Carlos. Madrid. Spain; Emilio Renes Carreño, MD, PhD, Principal Investigator — Hospital Universitario 12 de Octubre. Madrid. Spain; María Lourdes Cordero Lorenzana, MD, Principal Investigator — Complejo Hospitalario Universitario A Coruña. Galicia. Spain.; Juan Carlos López Delgado, MD, PhD, Principal Investigator — Hospital Universitario de Bellvitge. Cataluña. Spain.; Paola Zárate Chug, MD, Principal Investigator — Hospital Universitario Miguel Servet. Zaragoza. Spain.; Belén Vila García, MD, Principal Investigator — Hospital Universitario Infanta Cristina. Parla. Madrid. Spain; Rosa María Gastaldo Simeón, MD, Principal Investigator — Hospital de Manacor. Mallorca. Islas Baleares. Spain; Fátima Martínez Lozano Aranaga, MD, Principal Investigator — Hospital General Universitario Reina Sofía. Murcia. Spain.; Carolina Lorencio Cárdenas, MD, Principal Investigator — Hospital Universitario de Girona Josep Trueta. Gerona. Spain; Mónica Zamora Elson, MD, Principal Investigator — Hospital de Barbastro. Huesca. Aragón. Spain.; Clara Vaquerizo Alonso, MD, Principal Investigator — Hospital Universitario de Fuenlabrada. Madrid. Spain.; María Luisa Bordejé Laguna, MD, Principal Investigator — Hospital Universitario Germans Trias i Pujol. Badalona. Barcelona. Cataluña. Spain.; Esther Portugal Rodríguez, MD, Principal Investigator — Hospital Universitario Lucus Augusti. Lugo. Galicia. Spain.; Lluís Servià Goixart, MD, PhD, Principal Investigator — Hospital Universitario Arnau de Villanova. Lérida. Cataluña. Spain.; Ana Martín Luengo, MD, Principal Investigator — Hospital Universitario Río Ortega. Valladolid. Castilla y León. Spain; Carmen Martín Parra, MD, Principal Investigator — Hospital Universitario del Tajo. Aranjuez. Madrid. Spain; Lidón Mateu Campos, MD, PhD, Principal Investigator — Hospital General Universitario de Castellón. Comunidad Valenciana. Spain; Juan Francisco Fernández Ortega, MD, Principal Investigator — Hospital Regional Universitario de Málaga. Andalucía. Spain; Carlos Serón Arbeloa, MD, PhD, Principal Investigator — Hospital de San Jorge. Huesca. Aragón. Spain; Elisabeth Navas Moya, MD, Principal Investigator — Hospital Universitario Mútua Terrassa. Barcelona. Spain.; María del Mar Juan Díaz, MD, Principal Investigator — Hospital Clínico Universitario de Valencia. Comunidad Valenciana. Spain; Alexander Agrifolio Rotaeche, MD, Principal Investigator — Hospital Universitario La Paz
Locations (23):
- Spain (23):
  - Hospital Regional Universitario de Málaga, Málaga, Andalusia
  - Hospital de San Jorge, Huesca, Aragon
  - Hospital de Barbastro, Huesca, Aragon
  - Hospital Universitario Miguel Servet, Zaragoza, Aragon
  - Hospital de Manacor., Palma de Mallorca, Balearic Islands
  - Hospital Universitario Río Hortega, Valladolid, Castille and León
  - Hospital Universitario de Bellvitge, Barcelona, Catalonia
  - Hospital Universitario Germans Trias i Pujol, Barcelona, Catalonia
  - Hospital Universitario de Girona Josep Trueta, Girona, Catalonia
  - Hospital Universitario Arnau de Villanova, Lleida, Catalonia
  - Hospital Universitario Mútua Terrassa, Terrassa, Catalonia
  - Complejo Hospitalario Universitario A Coruña, A Coruña, Galicia
  - Hospital Universitario Lucus Augusti, Lugo, Galicia
  - Hospital Universitario del Tajo, Aranjuez, Madrid
  - Hospital Universitario de Fuenlabrada, Fuenlabrada, Madrid
  - Hospital Universitario Severo Ochoa, Leganés, Madrid
  - Hospital Universitario Infanta Cristina, Parla, Madrid
  - Hospital General Universitario de Castellón, Castellon, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital General Universitario Reina Sofía, Murcia

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and Informed Consent Form would be shared with other researchers
Supporting Information: Study Protocol, ICF
Time Frame: From January 2018 to December 2018.
Access Criteria: Contact with Dr. Flordelís Lasierra (email: makalyconru@hotmail.com).